CLINICAL TRIAL: NCT06283069
Title: Relationship Between Lifestyle Indicators (Healthy Behaviours) and Cardiovascular Clinical Parameters (Healthy Factors)
Brief Title: Relationship Between Lifestyle Indicators and Cardiovascular Clinical Parameters
Acronym: RICH
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 45C301
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases; Lifestyle; Nutrition, Healthy; Physical Inactivity; Stress; Sleep
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: compilation of a questionnaire about LifeStyle — compilation of a questionnaire about LifeStyle

SUMMARY:
The goal of the study is to build a Register accruing data derived from the compilation of the questionnaire about LifeStyle for a population both of adults and of young boys and girls. The investigators are confident that in this way they will be able to expand the database they already have. The investigators will be able to increase the strength of the correlations between LS indices and health indicators. In particular, the investigators will emphasize the relationship between physical activity, stress, and diet quality on one hand, and on the other, they will focus on physiological parameters, like arterial pressure, gluco-lipid profile, and possible pathologies.

ELIGIBILITY:
Inclusion Criteria:

- ability to provide informed consent in compliance with the rules of Good Clinical Practice and current national regulations

Exclusion Criteria:

* inability to fill in the questionnaire
* inability to provide informed consent
* unwillingness to participate in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants / patients (both adults and children from 6 years of age) who are referred by their General Practitioner to the Exercise Medicine Unit of the IRCCS Istituto Auxologico Italiano for an internal medicine visit, or other clinical examinations such as evaluation of the autonomic nervous system through spectral analysis of the variability of cardiovascular parameters, or bioimpedance analysis.
  Only those persons who voluntarily provide their consent will participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2033-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
weekly physical activity volume | through study completion, an average of 1 year
  short version of International Physical Activity Questionnaire, which focuses on intensity (nominally estimated in Metabolic Equivalents - MET - according to the type of activity) and duration (in minutes) of physical activity. The following levels will be considered: brisk walking (≈ 3.3 METs), other modalities of activity of moderate intensity (≈ 4.0 METs), and activities of vigorous intensity (≈ 8.0 METs)

SECONDARY OUTCOMES:
nutrition quality | through study completion, an average of 1 year
  American Heart Association (AHA) Diet Score
weight | through study completion, an average of 1 year
  kg
height | through study completion, an average of 1 year
  cm
blood pressure | through study completion, an average of 1 year
  mmHg
perception of stress, fatigue, and somatic symptoms | through study completion, an average of 1 year
  short version of 4SQ questionnaire considering 4 specific symptoms (total score ranging from 0 to 40)
glycemia | through study completion, an average of 1 year
  mg/dl
cholesterol | through study completion, an average of 1 year
  mg/dl
creatinine | through study completion, an average of 1 year
  mg/dl
waist circumference | through study completion, an average of 1 year
  cm
heart rate | through study completion, an average of 1 year
  bpm

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy